CLINICAL TRIAL: NCT02720107
Title: Long-term Follow up of Patients With Relapsing-remitting Multiple Sclerosis Enrolled in the Multicenter, Single-arm, Open-label Biobank Study (CFTY720DDE01), to Investigate Changes in Biomarkers After 48 Months of Treatment With 0.5 mg Fingolimod (FTY720)
Brief Title: Follow up Study of Patients on Fingolimod Who Were Enrolled in the Original Biobank Study (CFTY720DDE01)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CFTY720DDE01E1
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: fingolimod; Biomarker; Multiple sclerosis; Relapsing-remitting multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fingolimod (Experimental): Patients did not receive any protocol specified treatment during this follow-up study. Patients remained on their current treatment regime (fingolimod), as determined by their regular treating physician (i.e. 0.5 mg fingolimod daily, single-arm).
  Interventions: Drug: fingolimod

INTERVENTIONS:
Drug: fingolimod

SUMMARY:
The purpose of this single visit extension study is to explore immune status in RRMS patients treated for at least 48 months with fingolimod. Long-term changes in T cell counts will be compared to short-term changes in immune status (baseline to month 6) after treatment start with fingolimod as assessed in the original Biobank study (CFTY720DDE01).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent before any assessment was performed.
2. Randomized in study CFTY720DDE01 and received at least one dose of study drug (fingolimod) and completed the study.
3. Continuous intake of fingolimod after end of study CFTY720DDE01 with a maximum treatment interruption of 3 months in total before entering this study.
4. Parallel participation at study CFTY720DDE02 (Pangaea NIS) was allowed.

Exclusion criteriat:

1. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human Chorionic Gonadotropin (hCG) laboratory test.
2. Patients with onset of an acute relapse had to postpone their evaluation until deemed stable from relapse by treating physician, but at least for 1 month since end of relapse.
3. Patients that received immunomodulating or immunosuppressive MS treatments other than fingolimod since completion of study CFTY720DDE01 as for example: Natalizumab,Alemtuzumab, Dimethyl fumarate, Teriflunomide, intravenous Immunoglobulins,Mitoxantrone, Methotrexate, Azathioprine or experimental immunomodulating-immunosuppressive therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- Germany (24):
  - Novartis Investigative Site, Ostfildern, Baden-Wurttemberg
  - Novartis Investigative Site, Altenholz-Stift, Germany
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Celle
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Klingenmünster
  - Novartis Investigative Site, Lappersdorf
  - Novartis Investigative Site, Leverkusen
  - Novartis Investigative Site, Mönchengladbach
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neuburg an der Donau
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Singen
  - Novartis Investigative Site, Troisdorf
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Unterhaching

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 133 patients enrolled in the study but only 130 received drug
Period: Overall Study
Arm/Group | Fingolimod
Started | 130
Completed | 130
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fingolimod
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 47
Multiple Sclerosis History at screening of CFTY720DDE01 (Core) [Mean (Standard Deviation); unit: years] — Difference in years between first symptoms of Multiple Sclerosis (MS)and diagnosis is calculated as date of diagnosis minus date of first symptoms Difference between diagnosis and treatment start in Core is calculated as date of first treatment in Core minus date of diagnosis.
  years
    Difference of first symptons and diagnosis | 2.4 (3.56)
    Difference of dagnosis and tx start in Core | 8.6 (6.23)

OUTCOME MEASURES:

1. Primary Outcome: Change in T Cells Status (Decrease or Increase) at Month 48 (FAS)
Description: Aim of trial was to was to show reduction of CD4+ and CD8+ naïve T cells (CCR7+CD45RA+), central memory T cells (CCR7+CD45RA-), central memory Th17 cells (CD4+ CCR4+ and CCR6+), and an elevation of 2 types of effector memory T cells TEM (CCR7- CD45RA-) and TEMRA (CCR7- CD45RA+) in peripheral venous blood. Changes from baseline to month 48 in biomarkers were analyzed for all patients in the FAS.
Time Frame: Baseline up to approximately 48 months
Population: required baseline and month 48 visit measurement of the respective cell count
Measure: Least Squares Mean (Standard Error); unit: percentage of parent population
Arm/Group | Fingolimod
Number analyzed (Participants) | 130
percentage of parent population
  CD4+ Naïve T cells: number analyzed (Participants) | 121
  CD4+ Naïve T cells | -23.7 (0.62)
  CD4+Central memory T cells: number analyzed (Participants) | 120
  CD4+Central memory T cells | -1.2 (0.59)
  CD4+ Effector memory T cells: number analyzed (Participants) | 121
  CD4+ Effector memory T cells | 22.2 (2.37)
  CD8+ Naïve T cells: number analyzed (Participants) | 121
  CD8+ Naïve T cells | -37.2 (0.38)
  CD8+ Central memory T cells: number analyzed (Participants) | 121
  CD8+ Central memory T cells | -1.6 (0.07)
  CD8+ Effector memory T cells: number analyzed (Participants) | 121
  CD8+ Effector memory T cells | -12.9 (1.59)
  TH17 central memory cells: number analyzed (Participants) | 35
  TH17 central memory cells | -0.6 (0.03)
Statistical Analysis 1: Comparison: Fingolimod; CD4+ Naïve T cells; Test type: Superiority or Other; p < 0.0001, ANCOVA — The ANCOVA model included the covariates center, baseline of corresponding cell counts from Core study, sex and duration of disease until start of Core study
Statistical Analysis 2: Comparison: Fingolimod; CD4+ Central memory T cells; Test type: Superiority or Other; p = 0.0493, ANCOVA — The ANCOVA model included the covariates center, baseline of corresponding cell counts from study Core study, sex and duration of disease until start of Core study
Statistical Analysis 3: Comparison: Fingolimod; CD4+ Effector memory T cells; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Fingolimod; CD8+ Naïve T cells; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Fingolimod; CD8+ Central memory T cells; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Fingolimod; CD8+ Effector memory T cells; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Fingolimod; TH17 central memory cells; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants With Disability Progression as Measured by Expanded Disability Status Scale (EDSS) (FAS)
Description: EDSS is a scale for assessing neurologic impairment in MS. It is a two-part system including
  (1) a series of scores in each of eight functional systems, and (2) the EDSS steps (ranging from 0 (normal) to 10 (death due to MS). The definition of disability progression was based on increases in EDSS from baseline and depended on the EDSS baseline value: Disability progression was defined as a 1.5 increase in EDSS from baseline in subjects with a baseline EDSS score between 0.0 and 0.5, as a 1.0 increase in EDSS from baseline in subjects with a baseline EDSS score between 1.0 and 5.0 inclusive and 0.5 increase from baseline in subjects with EDSS score > 5.0.
Time Frame: Baseline up to approximately 48 months
Measure: Number; unit: percentage of participants
Arm/Group | Fingolimod
Number analyzed (Participants) | 130
percentage of participants | 21.54

3. Secondary Outcome: Change From Baseline in Disability Progression Assessed With the Expanded Disability Status Scale (EDSS) at Month 6 and Month 48 (FAS)
Description: as for outcome 2
Time Frame: Baseline, month 6 up to approximately 48 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fingolimod
Number analyzed (Participants) | 130
scores on a scale
  Baseline | 2.7 (1.17)
  Month 6 | 2.6 (1.38)
  Month 48 | 2.7 (1.52)
  Change from baseline to month 6 | -0.1 (0.69)
  Change from month 6 to month 48 | 0.2 (1.18)
  Change from baseline to month 48 | 0.0 (1.19)

4. Secondary Outcome: Change in Immune Status of B Cells, Monocytes and Natural Killer Cells (NK) Cells (FAS)
Description: Changes in immune status of B cells (CD19+, CD20+, CD69+), monocytes (CD14+) and NK cells (CD56+) were analyzed as a percentage of parent cell population (CD4+, CD8+ or total lymphocytes) by flow cytometry
Time Frame: Baseline up to approximately 48 months
Population: analysis required valid samples for baseline and month 48
Measure: Least Squares Mean (Standard Error); unit: percentage of parent population
Arm/Group | Fingolimod
Number analyzed (Participants) | 130
percentage of parent population
  B cells: number analyzed (Participants) | 95
  B cells | -7.2 (0.42)
  Monocytes: number analyzed (Participants) | 95
  Monocytes | 42.3 (2.03)
  Natural Killer cells: number analyzed (Participants) | 82
  Natural Killer cells | 28.0 (2.09)

ADVERSE EVENTS:
Time Frame: (Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.(approximately 48 months)
Groups:
- Fingolimod 0.5 mg: fingolimod 0.5 mg
Arm/Group | Fingolimod 0.5 mg
Serious Adverse Events (participants affected / at risk) | 0/130
Other Adverse Events (participants affected / at risk) | 1/130
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 0.5 mg (N=130)
Blood immunoglobulin M decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.